CLINICAL TRIAL: NCT02703623
Title: A Dynamic Allocation Modular Sequential Trial of Approved and Promising Therapies in Men With Metastatic Castrate Resistant Prostate Cancer
Brief Title: Abiraterone Acetate, Prednisone, and Apalutamide With or Without Ipilimumab or Cabazitaxel and Carboplatin in Treating Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0386; NCI-2016-00670 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2014-0386 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Castration Levels of Testosterone; Castration-Resistant Prostate Carcinoma; Metastatic Prostate Carcinoma; PSA Progression; Stage IV Prostate Adenocarcinoma AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; apalutamide; cabazitaxel; XRP6258; Carboplatin; Ipilimumab; CTLA-4 Antigen; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 2A (abiraterone acetate, prednisone, apalutamide) (Experimental): Patients receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Other: Laboratory Biomarker Analysis; Drug: Prednisone
- Arm 2B (abiraterone acetate, prednisone, ARN-509, ipilimumab) (Experimental): Patients receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily. Patients also receive ipilimumab IV over 90 minutes on day 1 of courses 4-7. Courses repeat every 3 weeks in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Biological: Ipilimumab; Other: Laboratory Biomarker Analysis; Drug: Prednisone
- Arm 3(abiraterone, prednisone, ARN509,cabazitaxel,carboplatin) (Active Comparator): Patients receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily. Patients also receive cabazitaxel IV over 60 minutes and carboplatin IV, over 60 minutes on day 1 of courses 4-13. Courses repeat every 3 weeks in the absence of disease progression or unexpected toxicity.
  Interventions: Drug: Abiraterone Acetate; Drug: Apalutamide; Drug: Cabazitaxel; Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone Acetate — Given PO
  Other Names: CB7630; Zytiga
Drug: Apalutamide — Given PO
  Other Names: ARN 509; ARN-509; ARN509; JNJ 56021927; JNJ-56021927
Drug: Cabazitaxel — Given IV
  Other Names: Jevtana; RPR-116258A; Taxoid XRP6258; XRP-6258
  Arms: Arm 3(abiraterone, prednisone, ARN509,cabazitaxel,carboplatin)
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm 3(abiraterone, prednisone, ARN509,cabazitaxel,carboplatin)
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Arm 2B (abiraterone acetate, prednisone, ARN-509, ipilimumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone

SUMMARY:
This randomized phase II trial studies the side effects and how well abiraterone acetate, prednisone, and apalutamide work with or without ipilimumab or cabazitaxel and carboplatin in treating patients with castration-resistant prostate cancer that has spread to other places in the body. Androgens can cause the growth of prostate cancer cells. Drugs, such as abiraterone acetate and apalutamide may lessen the amount of androgens made by the body. Immunotherapy with monoclonal antibodies, such as ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as prednisone, cabazitaxel, and carboplatin work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. It is not yet known whether giving abiraterone acetate, prednisone, and apalutamide with or without ipilimumab or cabazitaxel and carboplatin may be a better way to treat patients with castration-resistant prostate cancer that has spread to other places in the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the overall survival (OS) of men with metastatic castration-resistant prostate cancer (mCRPC) who have SATISFACTORY features after to 8 weeks of maximal androgen receptor (AR)-inhibitory therapy and receive treatment with abiraterone acetate, prednisone and apalutamide plus or minus ipilimumab.

II. To estimate the OS of men with mCRPC who have UNSATISFACTORY features after to up to 8 weeks of maximal androgen receptor (AR)-inhibitory therapy and receive treatment with abiraterone acetate, prednisone, apalutamide, cabazitaxel and carboplatin.

III. To determine the TOXICITY PROFILE of the following combinations in men with mCRPC:

IIIa. Abiraterone acetate, prednisone, apalutamide. IIIb. Abiraterone acetate, prednisone, apalutamide and ipilimumab. IIIc. Abiraterone acetate, prednisone, apalutamide, cabazitaxel and carboplatin.

IV. To determine whether the BASELINE "AR RESPONSE SIGNATURE" correlates with SATISFACTORY or UNSATISFACTORY features after up to 8-weeks of treatment with abiraterone, prednisone and apalutamide.

SECONDARY OBJECTIVES:

I. To "pick the winner" in terms of time to treatment failure (TTF) between the following two combinations, in men with mCRPC and satisfactory features after 8 weeks of maximal AR-inhibitory therapy:

Ia. Abiraterone acetate, prednisone, apalutamide. Ib. Abiraterone acetate, prednisone, apalutamide and ipilimumab. II. To determine the TTF in men with mCRPC and unsatisfactory features after up to 8 weeks of maximal AR-inhibitory therapy ted with abiraterone acetate, prednisone, apalutamide, cabazitaxel and carboplatin.

III. To determine whether the "baseline AR response signature" predicts for benefit by prognostic grouping (satisfactory/unsatisfactory) and treatment arm.

IV. To investigate therapy-specific marker signatures (immune based, bone based and anaplastic) and their link to outcome.

V. To collect and archive bone marrow biopsy, bone marrow aspirate, serum, plasma, and tissue samples in study patients for later hypothesis generating associations.

OUTLINE: After an 8-week lead-in phase, patients with satisfactory decline in serum markers are randomized to 1 of 2 arms (Arm 2A or 2B), and patients with unsatisfactory decline in serum markers are assigned to Arm 3.

LEAD-IN PHASE: Patients receive abiraterone acetate orally (PO) daily, prednisone PO twice daily (BID), and apalutamide PO daily for 8 weeks in the absence of disease progression or unexpected toxicity.

ARM 2A: Patients receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily in the absence of disease progression or unexpected toxicity.

ARM 2B: Patients receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily. Patients also receive ipilimumab intravenously (IV) over 90 minutes on day 1 of courses 4-7. Courses repeat every 3 weeks in the absence of disease progression or unexpected toxicity.

ARM 3: Patients receive abiraterone acetate PO daily, prednisone PO BID, and apalutamide PO daily. Patients also receive cabazitaxel IV over 60 minutes and carboplatin IV over 60 minutes on day 1 of courses 4-13. Courses repeat every 3 weeks in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up at 14 and 30 days, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet the following criteria to be enrolled in this study:

1. Willing and able to provide written informed consent.
2. Male aged 18 years and above.
3. Histologically or cytologically confirmed adenocarcinoma of the prostate.
4. Presence of metastatic disease documented on imaging studies (bone scan, CT and/or MRI scans).
5. Patients must have documented evidence of progressive disease as defined by any of the following: a) PSA progression: minimum of 2 rising values (3 measurements) obtained a minimum of 7 days apart with the last result being at least >/= 1.0 ng/mL; b) New or increasing non-bone disease (RECIST 1.1 criteria); c) Positive bone scan with 2 or more new lesions (PCWG3).
6. Surgically or ongoing medically castrated, with baseline testosterone levels of ≤ 50 ng/dL (≤ 2.0 nM).
7. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
8. Hemoglobin ≥ 7.5 g/dL in the presence of bone marrow involvement independent of transfusion and/or growth factors within 3 months prior to enrollment.
9. Platelet count ≥100,000/μL independent of transfusion and/or growth factors within 3 months prior to enrollment.
10. Serum albumin ≥3.0g/dL.
11. Medications known to lower the seizure threshold (see Appendix H under prohibited medications) must be discontinued or substituted at least 4 weeks prior to study entry.
12. Absolute neutrophil count (ANC) ≥ 1,500/mm3
13. Calculated creatinine clearance (Cockcroft-Gault Equation) ≥ 40 mL/min.
14. Serum potassium ≥ Institutional Lower Limit of Normal (ILLN).
15. Serum magnesium ≥ ILLN.
16. Serum bilirubin < 1.5 x Institutional Upper Limit of Normal (IULN) (except for patients with known Gilbert's disease).
17. Serum AST or ALT < 2.5 x IULN for patients without liver metastases. For patients with liver metastases AST or ALT < 5 x IULN is allowed.
18. Able to swallow study drugs whole as a tablet/capsule.
19. Male subject with a female partner of childbearing potential or pregnant must agree to use two acceptable methods of contraception and not to donate sperm from time of Screening until 3 months after the last dose of study treatments as per Section 5.7. Patients must agree to tissue collection for correlative studies (including participation in PA13-0291 and PA13-0247 for MD Anderson participants) at the specified timepoints. (Additional details in Section 5.5.1.1).

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study:

Prior or Concurrent Treatments:

1. Any prior treatment with:

   * Ipilimumab
2. Treatment within 28 days of Cycle1 Day1:

   * Any other systemic therapy for prostate cancer (with the exception of LHRH agonists and LHRH antagonists for testosterone suppression Sipuleucel-T, and bisphosphonates and RANK-ligand inhibitors for bone metastases which are allowed).
   * Any other investigational product.
   * Any medications listed in Appendix H
3. Treatment within 12 months of Cycle 1 Day 1 with any Cyp17-lyase inhibitor, any 2 nd generation AR antagonist (e.g. enzalutamide), cabazitaxel orcarboplatin.
4. Patients treated with any Cyp17-lyase inhibitor, any 2nd generation AR antagonist (e.g. enzalutamide), cabazitaxel or carboplatin whose disease progressed while on treatment or within 3 months of its discontinuation. (Patients who have received any of these treatments more than 12 months from study entry and whose disease did not progress while on treatment or within 3 months of its discontinuation are allowed on study).
5. Patients whose disease is refractory (defined as evidence of disease progression while on drug or within 3 months of its discontinuation) to more than 2 lines of chemotherapy. Any number of chemotherapies to which the patient's disease is not refractory are allowed, as long as time on treatment did not exceed 6 months (counted from day 1 of cycle 1 to day 1 of the last cycle of treatment).
6. Flutamide (Eulexin) treatment within 4 weeks of Cycle 1, Day 1 and Bicalutamide (Casodex) or nilutamide (Nilandron) within 6 weeks of Cycle 1 Day 1 Exceptions: if progression is documented prior to this time interval, or if patient is deemed by the treating physician to be highly unlikely to respond to AR inhibitor withdrawal (e.g. if PSA did not decline for ≥3 months in response to AR inhibitor given as a second line or later intervention, or if patient has symptoms attributable to disease progression) only a 3 day washout prior to Cycle 1, Day 1 will be required for any of them.
7. Radiation therapy for treatment of the primary tumor within 6 weeks of Cycle 1, Day 1. Patients who have received palliative radiation and recovered areeligible.
8. Any chronic medical condition requiring a higher dose of corticosteroid than 10mg prednisone/prednisolone daily. Use of inhaled, intranasal, intra-articular and topical steroids are acceptable, as is a short course (i.e. ≤ 1 day) of corticosteroids to prevent a reaction to the IV contrast used for CT scans.

   Concurrent illnesses:
9. Active infection (requiring oral or IV antibiotics or antiviral therapy) or other medical condition that would make prednisone/prednisolone (corticosteroid) use contraindicated. Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. A malignancy [other than the one treated in this study] which required radiotherapy or systemic treatment within the past 5 years, or has a ≥ 30% probability of recurrence within 24 months (except for non-melanoma skin cancer or Ta urothelial carcinomas).
11. Uncontrolled hypertension (systolic BP ≥ 140 mmHg or diastolic BP ≥ 90 mmHg). Patients with a history of hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
12. Prolonged QTc interval on pre-entry electrocardiogram (≥ 450 msec).
13. Known active or symptomatic viral hepatitis or chronic liver disease.
14. Clinically significant heart disease as evidenced by myocardial infarction, or arterial thrombotic events in the past 6 months, severe or unstable angina, history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsade de pointes), New York Heart Association (NYHA) Class III-IV heart disease or cardiac ejection fraction measurement of < 40% at baseline.
15. Autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic progressive sclerosis [scleroderma and variants], Systemic Lupus Erythematosus, autoimmune vasculitis [e.g., Wegener's Granulomatosis] or autoimmune neuropathies (such as Guillain-Barre syndrome) are excluded from this study. Vitiligo and adequately controlled endocrine deficiencies such as hypothyroidism are not exclusionary.
16. Patients who have had a history of illness which put them at current risk for bowel perforation such as acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis.
17. History of seizure or known condition that may pre-dispose to seizure (including but not limited to prior stroke or loss of consciousness within 1 year prior to randomization, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing edema or mass effect).
18. Gastrointestinal disorder affecting absorption. Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events.
19. Untreated symptomatic spinal cord compressions.

    Other:
20. Prisoners or subjects who are involuntarily incarcerated.
21. Subjects who are compulsorily detained for treatment of either a psychiatric or physical (e.g. infectious disease) illness.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2016-05-18 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Up to 4 years
  Will be reported for each arm. Estimated by Bayesian posterior estimates along with the 95% credible intervals and presented using Kaplan-Meier curves.
Incidence of adverse events as measured by the method of Thall et al | Up to 4 years
  Will be reported overall as well as by grade and attribution to study drug for each arm.
Androgen receptor (AR) response marker signature | At baseline
  Chi-Square tests or chi-square exact tests at a two-sided significance level of 0.05 will be used to evaluate the association between "AR-response marker signatures" (good/bad) and the "allocation serum marker decline" (satisfactory/unsatisfactory).
Allocation serum marker decline | At 8 weeks
  Serum levels of prostate specific antigen (PSA) and circulating tumor cells (CTCs) will be evaluated and correlated with AR response marker signatures. Chi-Square tests or chi-square exact tests at a two-sided significance level of 0.05 will be used to evaluate the association between "AR-response marker signatures" (good/bad) and the "allocation serum marker decline" (satisfactory/unsatisfactory). Multivariate logistic regression analysis adjusting for the effects of other baseline factors will also be used to identify factors associated with a satisfactory allocation serum marker profile.

SECONDARY OUTCOMES:
Time to treatment failure (TTF) | Up to 4 years
  Estimated by Bayesian posterior estimates along with the 95% credible intervals and presented using Kaplan-Meier curves.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Aparicio, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson in Katy, Houston, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org